CLINICAL TRIAL: NCT03802435
Title: Comparison of Long-term Effect in Different Sessions of Perineural Injection With Dextrose for Carpal Tunnel Syndrome
Brief Title: Different Sessions of Perineural Injection With Dextrose for Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Yung-Tsan Wu, Attending Physician of Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Different PIT for CTS
Record Dates: First submitted 2019-01-09; First posted 2019-01-14 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Carpal Tunnel Syndrome
Keywords: perineural injection therapy; nerve hydrodissection
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Two-sessions of ultrasound-guided PIT (Experimental): two-sessions of ultrasound-guided PIT with 10cc 5% dextrose (3 months interval)
  Interventions: Procedure: two-sessions of ultrasound-guided PIT
- One-session of ultrasound-guided PIT (Active Comparator): one-session of ultrasound-guided PIT with 10cc 5% dextrose and 10cc normal saline separately (3 months interval)
  Interventions: Procedure: One-sessions of ultrasound-guided PIT
- Two-session of ultrasound-guided nerve hydrodissection (Placebo Comparator): two-sessions of ultrasound-guided PIT with nerve hydrodissection with 10cc normal saline (3 months interval).
  Interventions: Procedure: Placebo ultrasound-guided injection with nerve hydrodissection

INTERVENTIONS:
Procedure: two-sessions of ultrasound-guided PIT — two-sessions of ultrasound-guided PIT with 10cc D5W (3 months interval)
  Arms: Two-sessions of ultrasound-guided PIT
Procedure: One-sessions of ultrasound-guided PIT — One-session of ultrasound-guided PIT with 10cc D5W and 10cc normal saline separately (3 months interval)
  Arms: One-session of ultrasound-guided PIT
Procedure: Placebo ultrasound-guided injection with nerve hydrodissection — Two-sessions of ultrasound-guided PIT with nerve hydrodissection with 10cc normal saline (3 months interval).
  Arms: Two-session of ultrasound-guided nerve hydrodissection

SUMMARY:
Carpal tunnel syndrome (CTS) is the most common peripheral entrapment neuropathy with involving compression of the median nerve in the carpal tunnel. The technique of perineural injection therapy (PIT) by using 5% dextrose (D5W) is now commonly used for peeling the nerve from surrounding soft tissue (called nerve hydrodissection), which may help antineurogenic inflammation, allow the impulse to pass, and rescue the nerve with ischemic damage. However, the evidence and reference of PIT and nerve hydrodissection are very seldom until our series researches since 2017. Moreover, our research revealed PIT with D5W is more beneficial than that of corticosteroid in patients with mild-to-moderate CTS at 4 to 6 months postinjection. However, the accumulative effect and long-term effect (more than 6 months) of PIT is still unknown. Hence, we design a randomized, double- blind, controlled trail to assess the long-term effect of ultrasound-guided PIT in patients with CTS. The aim one is to survey the possible accumulative effect of different sessions of PIT (6 months follow-up) and aim two is to evaluate the long-term effect and safety of PIT (one year follow-up).

DETAILED DESCRIPTION:
After obtaining written informed consent, patients clinically diagnosed with mild-to-moderate CTS were includes and randomized into three groups. Group A, patients received two-sessions of ultrasound-guided PIT with 10cc D5W (3 months interval); Group B, patients received one-session of ultrasound-guided PIT with 10cc D5W and 5cc normal saline separately (3 months interval); Group C (control group), patients received two-sessions of ultrasound-guided PIT with nerve hydrodissection with 10cc normal saline. The primary outcome is Boston Carpal Tunnel Syndrome Questionnaire (BCTQ) and secondary outcomes include visual analog scale (VAS), cross-sectional area (CSA) of the median nerve, nerve conduction velocity of the median nerve, and Global assessment of treatment. The evaluations were performed pretreatment as well as on the 1st, 3rd, 6th, 9th month and one year after first injection.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-80 year-old.
* Diagnosis was confirmed using an electrophysiological study

Exclusion Criteria:

* Cancer
* Coagulopathy
* Pregnancy
* Inflammation status
* Cervical radiculopathy
* Polyneuropathy, brachial plexopathy
* Thoracic outlet syndrome
* Previously undergone wrist surgery or steroid injection for CTS

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline of severity of symptoms and functional status on 1st, 3rd, 6th, 9th month and one year after injection | Pre-treatment, 1st, 3rd, 6th, 9th month and one year after injection
  Boston carpal tunnel syndrome questionnaire (BCTQ) is a frequently used patient-based questionnaire for measurement of CTS which encompasses two components. In total, 11 questions and 8 items were evaluated to rate the symptom severity scale (SSS) and functional status scale (FSS), respectively. Both subscales range from 1 to 5 with a higher score indicating a higher degree of disability. The mean of total SSS and FSS divided with each item score were used for further analysis.

SECONDARY OUTCOMES:
Change from baseline of pain on 1st, 3rd, 6th, 9th month and one year after injection | Pre-treatment, 1st, 3rd, 6th, 9th month and one year after injection
  Digital pain severity or paresthesia/dysthesia was evaluated using visual analog scale (VAS). Pain score scale ranged from 0 to 10, with 10 indicating the most severe pain.
Change from baseline of cross-sectional area of the median nerve on 1st, 3rd, 6th, 9th month and one year after injection | Pre-treatment, 1st, 3rd, 6th, 9th month and one year after injection
  Using the musculoskeletal sonogram to measure the cross-sectional area of the median nerve before treatment and multiple time frame after treatment.
Change from baseline of electrophysiological measurement on 1st, 3rd, 6th, 9th month and one year after injection | Pre-treatment, 1st, 3rd, 6th, 9th month and one year after injection
  Antidromic sensory nerve conduction velocity of the median nerve before treatment and multiple time frame after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Tsan Wu, MD, Principal Investigator — Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital
Locations (1):
- Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital, Taipei, Neihu District, Taiwan

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Wu YT, Chen SR, Li TY, Ho TY, Shen YP, Tsai CK, Chen LC. Nerve hydrodissection for carpal tunnel syndrome: A prospective, randomized, double-blind, controlled trial. Muscle Nerve. 2019 Feb;59(2):174-180. doi: 10.1002/mus.26358. Epub 2018 Dec 4. PMID 30339737
- [Result] Wu YT, Ho TY, Chou YC, Ke MJ, Li TY, Tsai CK, Chen LC. Six-month Efficacy of Perineural Dextrose for Carpal Tunnel Syndrome: A Prospective, Randomized, Double-Blind, Controlled Trial. Mayo Clin Proc. 2017 Aug;92(8):1179-1189. doi: 10.1016/j.mayocp.2017.05.025. PMID 28778254
- [Result] Wu YT, Ke MJ, Ho TY, Li TY, Shen YP, Chen LC. Randomized double-blinded clinical trial of 5% dextrose versus triamcinolone injection for carpal tunnel syndrome patients. Ann Neurol. 2018 Oct;84(4):601-610. doi: 10.1002/ana.25332. Epub 2018 Oct 4. PMID 30187524